CLINICAL TRIAL: NCT04702659
Title: The Study of Clinical Observation About Chinese Medicine Zhengyi Prescription
Brief Title: Chinese Medicine Zhengyi Prescription Tea Bag
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-10-002B
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Herbal Interaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chinese herbal tea bags can adjust physiological functions, help protect power, and give positive energy to the body. This prescription not only focuses on regulating the patient's physical function, but also helps to enhance physical strength.

DETAILED DESCRIPTION:
In Taiwan ,acoording to the TCM theories and viewpoints, Chinese herbal medicine plays an important role in clinical drug application.TCM compound combinations for different diseases, emphasizing the complementarity and balance of ingredients, natural gentleness, uniqueness and efficacy are widely accepted by the public.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 20, those who have no chronic respiratory disease or those who have been diagnosed as nasal and sinusitis by a doctor, whose clinical diagnosis includes subjects with allergic rhinitis.

Exclusion Criteria:

1. Patient characteristics: age, gender, weight, education level, race, pregnancy and breastfeeding status, smoking, drinking, caffeine, alcohol or drug poisoning, diet and nutritional status, physical limitations, genetic history, etc. Exclude women under the age of 20, unable to order their behavior, pregnant or breast-feeding women
2. Disease characteristics: Subjects who have been diagnosis of mental illness by doctors, as well as long-term diarrhea or long-term use of Chinese medicine.
3. Environmental characteristics: other conditions that make patients unable to cooperate. Such as unsuitability after screening, not signing the subject consent form, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants have no chronic respiratory disease or those who have been diagnosed as nasal and sinusitis by a doctor, whose clinical diagnosis includes subjects with allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
questionnaire-the Chinese Version of the 31-Item Rhinosinusitis Outcome Measure | 28days
  The questionnaire contains a total of 31 assessment items:
  Divided into 7 major aspects: nasal symptoms (6 questions), eye symptoms (2 questions), Sleep condition (4 questions), ear symptoms (5 questions), overall symptoms (7 questions), daily life Influence (4 questions) and the influence of emotions (3 questions). According to the patient's four weeks,the symptoms within are scored for each item, and the first category is to evaluate the symptoms of this item. The first score ranges from 0 points (no such symptoms) to 5 points (extremely severe Heavy); The second category is to assess the importance of this symptom to the patient, starting from 1 Points (not important) to 4 points (very important). Multiply these two fractions together to get the symptom-impact score , this is the individual evaluation score of each patient for each symptom.

CONTACTS AND LOCATIONS:
Overall Officials: chang kaiwei, master, Principal Investigator — TaipeiVGH Center for Traditional Medicine
Locations (1):
- Center for Traditional Medicine, Taipei Veterans General Hospital, Taipei, Taiwan